CLINICAL TRIAL: NCT03681457
Title: A Phase 1, Open-label, Single-dose, Multi-center, Parallel Group Study to Evaluate the Pharmacokinetics of Tropifexor (LJN452) in Subjects With Mild, Moderate or Severe Hepatic Impairment Compared to Healthy Control Subjects
Brief Title: Evaluation of the Pharmacokinetics of Tropifexor in Subjects With Mild, Moderate, or Severe Hepatic Impairment Compared to Healthy Control Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLJN452A2109
Record Dates: First submitted 2018-09-11; First posted 2018-09-24 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-09

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: LJN452; tropifexor; PK; safety; healthy subjects; hepatically impaired; Nonalcoholic Steatohepatitis; Nonalcoholic Fatty Liver Disease; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — tropifexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 - Normal Hepatic Function (Other): Normal hepatic function - Control - control group
  Interventions: Drug: LJN452
- Group 2 - Mild Hepatic Impairment (Experimental): Mild hepatic impairment - Child-Pugh A (Score 5-6)
  Interventions: Drug: LJN452
- Group 3 - Moderate Hepatic Impairment (Experimental): Moderate hepatic impairment - Child-Pugh B (Score 7-9)
  Interventions: Drug: LJN452
- Group 4 - Severe Hepatic Impairment (Experimental): Severe hepatic impairment - Child-Pugh C (score 10-15)
  Interventions: Drug: LJN452

INTERVENTIONS:
Drug: LJN452 — Dose A single dose

SUMMARY:
The primary purpose of this study is to evaluate the effect of hepatic impairment on the systemic exposure of tropifexor and to evaluate the safety of tropifexor in subjects with hepatic impairment. The results of this study will support treatment and dosing decisions for patients with varying degrees of hepatic impairment.

ELIGIBILITY:
All subjects:

Inclusions Criteria:

* Subjects must weight at least 50 kg, with a BMI within the range of 18 to 38 kg/m2
* Must be willing to remain in the clinical research unit as required by the protocol

Exclusion Criteria:

* Use of other study drugs at the time of enrollment, or within 5 half-lives of enrollment, or within 30 days, whichever is longer; or longer if required by local regulations
* History of hypersensitivity to the study treatment or to drugs of similar chemical classes
* Pregnant or nursing women
* Women of child-bearing potential

Healthy Volunteers:

Inclusion Criteria:

- In good health as determined by past medical history, physical examination, ECG, laboratory tests, and urinalysis at Screening.

Exclusion Criteria:

* Liver disease or liver injury
* Chronic infection with Hepatitis B or Hepatitis C
* History or presence of impaired renal function

Hepatically Impaired Subjects:

Inclusion Criteria:

- Hepatic impairment as defined by the Child-Pugh classification for severity of liver disease

Exclusion Criteria:

* Severe complications of liver disease within the preceding 3 months
* Emergency room visit or hospitalization due to liver disease within the preceding 3 months for mildly and moderately hepatically impaired subjects, and within the preceding 1 month for severely hepatically impaired subjects
* Subject has received liver transplant at any time in the past and is on immunosuppressant therapy
* Acute Hepatitis B or Hepatitis C infection

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Cmax | Up to 8 days
  The maximum (peak) observed drug concentration after single dose administration (mass x volume-1)
Tmax | Up to 8 days
  Time to reach the maximum (peak) plasma drug concentration after single dose administration (time)
AUClast | Up to 8 days
  The area under the concentration-time curve from time zero to the time of the last quantifiable concentration sampling time (mass x time x volume-1)
AUCinf | Up to 8 days
  The area under the concentration-time curve from time zero to infinity (mass x time x volume-1)
T1/2 | Up to 8 days
  The elimination half-life associated with the terminal slope of a semi-logarithmic concentration-time curve
CL/F | Up to 8 days
  The apparent total body clearance of the drug from plasma (volume x time-1)
Vz/F | Up to 8 days
  The apparent volume of distribution during the terminal phase

SECONDARY OUTCOMES:
fu | Day 1
  Fraction of analyte unbound calculated in-vitro
Cmax,u | Day 1
  The maximum (peak) observed plasma drug concentration after single dose administration (Cmax) of unbound drug (mass x time x volume-1), calculated as Cmax*fu
AUClast,u | Day 1
  The area under the concentration-time curve from time zero to the last quantifiable concentration sampling time of unbound drug (mass x time x volume-1), calculated as AUClast*fu
AUCinf,u | Day 1
  The area under the concentration-time curve from time zero to infinity of unbound drug (mass x time x volume-1), calculated as AUCinf*fu
CL/F,u | Day 1
  The apparent total body clearance of drug from the plasma of unbound drug (volume x time-1), calculated as CL/F/fu

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CCLJN452A2109 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17722
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=555